CLINICAL TRIAL: NCT01043588
Title: Transurethral Resection of the Prostate With Photo Selective Vaporization of the Prostate Using the High Powered 532nm Laser Obstructive Benign Prostatic Hyperplasia Management: Focus on Efficiency and Cost-effectiveness
Brief Title: TRP Versus Photo Selective Vaporization for Obstructive Benign Prostatic Hyperplasia Management
Acronym: REVAPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); American Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K060401
Record Dates: First submitted 2009-12-21; First posted 2010-01-07 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2012-12

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Surgery; Prostate; Laser 532 nm; Photo selective Vaporization of the Prostate (PVP); TransUrethral Resection of the Prostate (TURP); Men health
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 : TURP (Other): Surgery: TransUrethral Resection of the Prostate
  Interventions: Procedure: TURP
- 2 : PVP (Other): Surgery: Photo selective Vaporization of the Prostate
  Interventions: Procedure: PVP

INTERVENTIONS:
Procedure: TURP — TransUrethral Resection of the Prostate
  Arms: 1 : TURP
Procedure: PVP — Photo selective Vaporization of the Prostate
  Arms: 2 : PVP

SUMMARY:
The aim of this study is to compare medical efficacy and cost effectiveness of two surgical options for obstructive BPH management : transurethral resection of the prostate with photo selective vaporization of the prostate using the high powered 532nm laser.

DETAILED DESCRIPTION:
The aim of this study is to compare medical efficacy and cost effectiveness of two surgical options for obstructive BPH management : transurethral resection of the prostate with photo selective vaporization of the prostate using the high powered 532nm laser. Patients were randomized in two groups after inclusion. Perioperative data were collected, and follow-up was conducted for one month.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 50 years of age or older.
2. American Society of Anesthesiology (ASA) classification of physical status, class 1-3
3. Signed an informed consent at the beginning of the study.
4. Patients presenting with LUTS associated to benign prostatic enlargement for more than 3 months, needing a surgical management, with at least one of the following situations: disability score ≥3, I-PSS ≥12, or full urinary retention
5. Qmax ≤12ml /s for no drained patients with voided volume> 125 ml.
6. Estimated prostate weight between 25g and 80g
7. Patient free of catheter with PVR ≤ 300cc
8. Patient without renal disorders.
9. No prostate cancer suspicion at clinical examination, including DRE.
10. PSA ≤ 10 ng/ml, with negative prostate biopsies of PSA is between 4 and 10 ng/mL if patient is 75 years or younger or has a life expectancy of more than 10 years.
11. In case of anticoagulation or anti-aggregation therapy, necessary preoperative visit by anaesthesiologist to determine the supply therapy around surgery.
12. In case of current BPH medical management, alpha blockers and herbal medicines should be stopped one week before surgery and 5-alpha-reductase-inhibitors should be stopped one month before surgery.
13. Patient must be affiliated to the French social healthcare or equivalent

Exclusion Criteria:

1. Uncontrolled cardiopulmonary disorder, previously or recently diagnosed by standard methods
2. Assessed sphincter detrusor dyssynergia, or myasthenia, multiple sclerosis, or Parkinson disease.
3. History of pelvic lesions with abdominal sphincter injury.
4. Urinary tract infection without antibiotics.
5. Patient with urinary catheter or suprapubic catheter because of an acute urinary retention linked to an alternative diagnosis or impaired bladder sensation.
6. Subject with neurogenic bladder and/or sphincter abnormalities
7. Subject with confirmed or suspected malignancy of the prostate or the bladder.
8. Previous prostatic surgery.
9. History of bladder stone, major hematuria, urethral stricture, bladder neck stenosis.
10. Patient having a prosthesis in the procedure area
11. Patient with an active anorectal disease
12. Treatment emergency
13. Individual unable to respect timing and visits determined by the protocol.
14. Constitutional hemostasis and coagulation abnormalities not linked to oral medications
15. Any disease or patient condition which can be a contra indication to his enrolment in the study, according to the investigator.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Hospital stay | end of hospitalization
Clinical symptoms at 1-yr follow-up evaluated with usual objective and subjective parameters | at one year

SECONDARY OUTCOMES:
Rate of complication needing re-hospitalisation or reintervention | from the surgical procedure until one year follow-up
Risk of ignoring a localized prostate cancer needing a curative management. | at one year
Total and post-operative costs during follow-up. | from the surgical procedure until one year follow-up
Evaluation of side effects during follow-up. | from the surgical procedure until one year follow-up
Patient satisfaction | during follow up
Evaluation of quality of life | during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand LUKACS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital TENON - Service d'Urologie, Paris, France

REFERENCES:
- [Background] Bachmann A, Schurch L, Ruszat R, Wyler SF, Seifert HH, Muller A, Lehmann K, Sulser T. Photoselective vaporization (PVP) versus transurethral resection of the prostate (TURP): a prospective bi-centre study of perioperative morbidity and early functional outcome. Eur Urol. 2005 Dec;48(6):965-71; discussion 972. doi: 10.1016/j.eururo.2005.07.001. Epub 2005 Jul 18. PMID 16126327
- [Derived] Lukacs B, Loeffler J, Bruyere F, Blanchet P, Gelet A, Coloby P, De la Taille A, Lemaire P, Baron JC, Cornu JN, Aout M, Rousseau H, Vicaut E; REVAPRO Study Group. Photoselective vaporization of the prostate with GreenLight 120-W laser compared with monopolar transurethral resection of the prostate: a multicenter randomized controlled trial. Eur Urol. 2012 Jun;61(6):1165-73. doi: 10.1016/j.eururo.2012.01.052. Epub 2012 Feb 8. PMID 22341632